CLINICAL TRIAL: NCT06756841
Title: A Single-arm Clinical Trial to Explore the Safety and Efficacy of Pulsed Electric Field (PEF) Therapy in Patients With Advanced or Unresectable Esophageal Squamous Cell Carcinoma
Brief Title: Safety and Efficacy Study of Pulsed Electric Field (PEF) Therapy in Patients With Advanced or Unresectable Esophageal Squamous Cell Carcinoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Energenx Medical LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC-001
Record Dates: First submitted 2024-12-09; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PEF treatment (Experimental): One group prospective clinical
  Interventions: Device: PEF treatment

INTERVENTIONS:
Device: PEF treatment — PEF energy delivery via endoscope

SUMMARY:
The goal of this clinical trial is to verify the safety and clinical benefit of pulsed electric field (PEF) treatment of advanced or unresectable esophageal squamous cell carcinoma patients.

The main questions it aims to answer are:

* Safety and feasibility of PEF treatment of patients with advanced or unresectable esophageal squamous cell carcinoma.
* Locoregional control of ablated lesions and quality of life assessment.
* Local and peripheral immunoregulation effect.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 20 years or older when signing the informed consent form.
2. Able to provide written informed consent, and understand and follow the study requirements and assessment schedule.
3. Screening period tumor patients ECOG performance status score of 0 or 1.
4. Laboratory test data within 7 days before the planned PEF treatment date during the screening period must meet the following standards.

   * Neutrophil count (ANC) ≥1500 cells/mm3
   * Platelet count ≥100,000 cells/mm3
   * Hemoglobin ≥9 g/dL or ≥5.6 mmol/L
   * Serum total bilirubin ≤ 1.5 x ULN.
5. Females of childbearing potential must have a negative serum pregnancy test at screening and be willing to undergo additional pregnancy testing during the study.

Exclusion Criteria:

1. Subjects with active respiratory tract infection who need antibiotic or antiviral treatment;
2. Patients with locally advanced ESCC whose tumors can be surgically removed by the investigator or can be potentially cured by radical chemoradiotherapy according to the judgment of local investigators.
3. Patients with esophageal lesions that severely invade adjacent organs (esophagus/bronchus or esophagus/aorta) and are assessed as high-risk esophageal leakage/fistula by the investigator.
4. Evidence of complete esophageal obstruction that is not suitable for treatment, and gastroscopy cannot be performed.
5. Patients with a history of esophageal stent implantation for esophageal obstruction;
6. Patients with a history of gastrointestinal bleeding in the past 4 weeks, or gastroscopy indicates a high risk of tumor ulcer bleeding.
7. Patients with obstruction caused by anastomotic stenosis without esophageal primary lesions after previous esophageal cancer surgery.
8. Patients with active leptomeningeal disease or brain metastasis.
9. Any active malignant tumor within 5 years before screening.
10. Subjects have undergone metal implantation surgery such as esophageal stents and airway stents. Or the patient has an implantable cardioverter-defibrillator, pacemaker or other implantable electronic device.
11. Patients with positive HIV test.
12. Subjects are currently participating in other research clinical trials;
13. Subjects who are considered by the investigator to have other high-risk conditions and are not suitable for gastroscopy and surgery;
14. Subjects who have adverse events that have not yet returned to baseline or stable levels due to previous anti-tumor treatment, except for adverse events that do not pose safety risks (such as hair loss and abnormal values of specific laboratory tests)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-12-25 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Safety of PEF treatment | 1 month
  evaluate the rate of AEs/SAEs associated with instrument-related/or surgical procedures within 30 days of PEF treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No